CLINICAL TRIAL: NCT00920647
Title: A Phase I/II, Randomized, Safety and Ascending Dose Ranging Study of Intrathecal Idursulfase-IT Administered in Conjunction With Intravenous Elaprase in Pediatric Patients With Hunter Syndrome and Cognitive Impairment
Brief Title: A Safety and Dose Ranging Study of Idursulfase (Intrathecal) Administration Via an Intrathecal Drug Delivery Device in Pediatric Patients With Hunter Syndrome Who Have Central Nervous System Involvement and Are Receiving Treatment With Elaprase®
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-HIT-045; 2010-020048-36 (EudraCT Number)
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Hunter Syndrome
Keywords: enlarged adenoids; hunters syndrome; enzyme replacement therapy; hunter's syndrome; mps society; Mucopolysaccharidosis (mps) 2; mps diagnosis; hunter disease; iduronate 2 sulfatase; idursulfase; hunters disease; hunter's syndrome treatment; mucopolysaccharides; hunter syndrome treatment; Mucopolysaccharidosis (mps) ii; elaprase; hunter syndrome therapy; lysosomal storage disease; hunter's disease; Mucopolysaccharidosis(MPS) II; Mucopolysaccharidosis(MPS)2; hunter's disease treatment; lysosomal storage disorder; chronic ear infection; mps symptoms; iduronate sulfatase; ert treatment
MeSH Terms: conditions — Mucopolysaccharidosis II; Mucopolysaccharidoses; Sudden Infant Death; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Other): Untreated Patients
  Interventions: Other: Control
- Idursulfase -IT (1 mg) (Experimental): monthly using an intrathecal drug delivery device (IDDD)
  Interventions: Drug: Idursulfase IT (1 mg)
- Idursulfase-IT (10 mg) (Experimental): monthly using an intrathecal drug delivery device (IDDD)
  Interventions: Drug: Idursulfase IT (10 mg)
- Idursulfase -IT (30 mg) (Experimental): monthly using an intrathecal drug delivery device (IDDD)
  Interventions: Drug: Idursulfase IT (30 mg)

INTERVENTIONS:
Other: Control — 3 dose cohorts were planned. Within each dose cohort, patients will be randomized to 1 of 2 treatment options: treatment with study drug or no treatment with 4 treated patients per dose group and a total of 4 untreated patients (1-2 untreated patients will be assigned in each dose cohort). They will not undergo surgical placement of an Intrathecal Drug Delivery Device (IDDD), and will not receive Idursulfase-IT.
  Arms: Control
Drug: Idursulfase IT (1 mg) — The original design of the study was to test the dose levels of 10, 30 and 100 mg. This was based on a calculation of a minimally effective dose around 10 mg, with subsequent dose levels being chosen as increasing half-log steps. During the conduct of the study; however, it became clear that the 10 mg dose elicited a strong Pharmacodynamic response, as measured by a dramatic and sustained drop in the CSF GAG levels. This indicated the need to explore a lower level as a minimally effective dose level, leading to the introduction of the 1 mg group. Enrollment of patients in this dose cohort will commence after the last patient has been enrolled in 30 mg dose cohort. 4 patients will be undergo surgical placement of an IDDD and receive 1 mg idursulfase-IT as an IT injection via an IDDD once per month (ie, every 28 days) for 6 month.
  Arms: Idursulfase -IT (1 mg)
Drug: Idursulfase IT (10 mg) — Patients will be enrolled in 10 mg dose cohort and 30 mg dose cohort in a sequential, escalating fashion. 4 patients will undergo surgical placement of an IDDD and receive 10 mg idursulfase-IT as an intrathecal (IT) injection via an IDDD once per month (ie, every 28 days) for 6 month.
  Arms: Idursulfase-IT (10 mg)
Drug: Idursulfase IT (30 mg) — Patients will be enrolled in 10 mg dose cohort and 30 mg dose cohort in a sequential, escalating fashion. 4 patients will undergo surgical placement of an IDDD and receive 30 mg idursulfase-IT as an IT injection via an IDDD once per month (ie, every 28 days) for 6 month.
  Arms: Idursulfase -IT (30 mg)

SUMMARY:
Elaprase (idursulfase), a large molecular protein, is not expected to cross the blood brain barrier at therapeutic levels when administered intravenously. A new formulation of idursulfase, idursulfase-IT, that differs from that of the intravenous (IV) formulation, Elaprase, has been developed to be suitable for delivery into the cerebrospinal fluid (CSF) via intrathecal administration.

This Phase I/II study is designed to obtain necessary safety and exposure data, as well as secondary and exploratory outcome measures, to be interpreted and used in the design of subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1a. A deficiency in iduronate-2-sulfatase enzyme activity of ≤10 % of the lower limit of the normal range as measured in plasma, fibroblasts, or leukocytes (based on normal range of measuring laboratory) AND

1b. A documented mutation in the iduronate-2-sulfatase gene OR A normal enzyme activity level of one other sulfatase as measured in plasma, fibroblasts, or leukocytes (based on normal range of measuring laboratory).

2. The patient is male and is ≥3 and <18 years of age .

3. The patient has evidence at Screening of early stage (duration and severity metrics per protocol) Hunter syndrome-related Central Nervous System (CNS) involvement, defined as:

* The patient has an Intelligence quotient (IQ) ≤77 OR
* There is evidence of a change of ≥1 but ≤2 standard deviations decline from a previous protocol-defined neurodevelopmental assessment. The duration of protocol-defined neurologic involvement is at least 3 months but less than 36 months as documented in the patient's medical history.

  4. The patient has received and tolerated a minimum of 6 months of treatment with weekly intravenous idursulfase, and has received 80% of the total planned infusions within that time frame, including having received 100% of the planned infusions within 4 weeks immediately preceding the surgical insertion of the IDDD.

  5. The patient must have sufficient auditory capacity, with or without aids, to complete the required protocol testing, and be compliant with wearing the aid on scheduled testing days.

  6. The patient, patient's parent(s), or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board / Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient. The guardians' consent must be obtained.

Exclusion Criteria:

1. The patient has clinically significant non-Hunter syndrome-related CNS involvement which is judged by the Investigator to be likely to interfere with the accurate administration and interpretation of protocol assessments.
2. The patient has an IQ ≥78
3. The patient has a CNS shunt.
4. The patient has experienced an infusion-related anaphylactoid event or has evidence of consistent severe adverse events related to treatment with Elaprase which, in the Investigator's opinion, may pose an unnecessary risk to the patient.
5. The patient has any known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptably high risk for anesthesia due to compromised airways or other conditions
6. The patient has a history of complications from previous lumbar punctures or technical challenges in conducting lumbar punctures such that the potential risks would exceed possible benefits for the patient.
7. The patient or patient's family has a history of neuroleptic malignant syndrome, malignant hyperthermia, or other anesthesia-related concerns.
8. The patient has a history of poorly controlled seizure disorder.
9. The patient has a significant medical or psychiatric comorbidity(ies) that might affect study data or confound the integrity of study results.
10. The patient is currently receiving chronic psychotropic therapy (e.g., neuroleptics, benzodiazepines, antidepressants, anticonvulsants, stimulants, etc.) which in the Investigator's opinion would likely affect the neurocognitive assessments. Intermittent use of selected short half-life agents (benzodiazepine, sedatives, etc.) may be permitted as long as there are 5 half-lives between last drug administered and study-related procedures including neurocognitive assessments.
11. The patient has received treatment with any investigational drug or device within the 30 days prior to study entry.
12. The patient has received a cord blood or bone marrow transplant at any time, or has received blood product transfusions within 90 days prior to Screening.
13. The patient is unable to comply with the protocol, (e.g., has significant hearing or vision impairment, a clinically relevant medical condition making implementation of the protocol difficult, unstable social situation, known clinically significant psychiatric/behavioral instability, is unable to return for safety evaluations, or is otherwise unlikely to complete the study), as determined by the Investigator.
14. The patient has skeletomuscular/spinal abnormalities or other contraindications for the surgical implantation of the IDDD.
15. The patient has an opening CSF pressure upon lumbar puncture that exceeds 30 cm H2O(water) .

Ages: 3 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2012-10-29 (Actual); Study Completion 2012-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Background] Muenzer J, Hendriksz CJ, Fan Z, Vijayaraghavan S, Perry V, Santra S, Solanki GA, Mascelli MA, Pan L, Wang N, Sciarappa K, Barbier AJ. A phase I/II study of intrathecal idursulfase-IT in children with severe mucopolysaccharidosis II. Genet Med. 2016 Jan;18(1):73-81. doi: 10.1038/gim.2015.36. Epub 2015 Apr 2. PMID 25834948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient enrolled on 18 November 2009. Patients were assigned randomly to active dose or no treatment. A total of 16 patients were randomized, 4 to each dose group and the no treatment arm.
Groups:
- Idursulfase IT (1 mg); Idursulfase IT (10 mg); Idursulfase IT (30 mg): monthly using an intrathecal drug delivery device (IDDD)
Period: Overall Study
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 4 | 4 | 16
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.64 (2.462) | 5.61 (1.799) | 4.34 (0.829) | 6.91 (1.678) | 6.38 (2.294)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 4 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 4 | 2 | 11
  United Kingdom | 1 | 2 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Event (SAE)
Time Frame: 6 months
Population: Abnormalities Any Time Post-baseline ITT Population
Measure: Number; unit: events
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
events | 0 | 8 | 3 | 3

2. Secondary Outcome: Change From Baseline in CSF Glycosaminoglycans [GAGs] at Week 27
Description: Percent Change from Baseline to Week 27
Time Frame: Baseline to Week 27
Measure: Mean (Standard Error); unit: % change
Groups:
- Control: Untreated Patients for 6 months, Observed Value
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
% change | 6.68 (6.301) | -79.03 (5.167) | -90.30 (2.917) | -88.87 (1.035)

3. Secondary Outcome: Level of Idursulfase in the CSF Compartment Resulting From Monthly Idursulfase IT Administrations
Description: Samples collected from patients treated at doses of 1 mg and 30 mg, as well as the control group, were below the lower limit of detection of the bioanalytical method (3.13 ng/mL)
Time Frame: Week 27 (end of study)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Idursulfase IT (1mg); Idursulfase IT (10 mg); Idursulfase IT (30 mg): monthly using an intrathecal drug delivery device (IDDD)
Arm/Group | Control | Idursulfase IT (1mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng/mL | NA (NA) — Samples collected from patients treated in the control group were below the lower limit of detection of the bioanalytical method (3.13 ng/mL). | NA (NA) — Samples collected from patients treated in the 1mg group were below the lower limit of detection of the bioanalytical method (3.13 ng/mL). | 6.74 (12.02) | NA (NA) — Samples collected from patients treated in the 30mg group were below the lower limit of detection of the bioanalytical method (3.13 ng/mL).

4. Primary Outcome: Number of Treatment Emergent Adverse Event (AE)
Description: ITT patient population
Time Frame: Baseline to week 23
Measure: Number; unit: events
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
events | 23 | 147 | 116 | 104

5. Primary Outcome: Safety Changes in Cerebrospinal Fluid (CSF)- White Blood Cells (WBC)
Description: White blood cell count in CSF was monitored throughout the study as a way of assessing any potential inflammation of the meninges induced by idursulfase-IT.
Time Frame: 6 months
Population: Abnormalities Any Time Post-baseline ITT Population
Measure: Number; unit: events
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
events | 0 | 3 | 1 | 2

6. Primary Outcome: Safety: Development of Anti-idursulfase Antibodies (CSF)
Description: Reflects development of anti-idursulfase antibodies post baseline.
Time Frame: 6 months
Population: Abnormalities Any Time Post-baseline ITT Population
Measure: Number; unit: participants
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
participants | 0 | 0 | 0 | 0

7. Primary Outcome: Safety: Development of Anti-idursulfase Antibodies (Serum)
Time Frame: 6 months
Population: Development of antibodies post Baseline-ITT Population
Measure: Number; unit: participants
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
participants | 1 | 0 | 0 | 0

8. Primary Outcome: Clinically Significant ECG Findings at Any Time During the Study.
Description: Electrocardiogram (ECG) parameters included: heart rate, sinus rhythm, atrial/ventricular hypertrophy, PR, QRS, QT and QTc intervals.
Time Frame: 6 months
Population: Abnormalities Any Time Post-baseline ITT Population
Measure: Number; unit: participants
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
participants | 0 | 0 | 1 | 0

9. Secondary Outcome: Concentration of Idursulfase in Serum After Single Administration (Week 3) in Conjunction With Elaprase
Description: Values below lower limit of quantitation (LLOQ) are listed as 0.
Time Frame: Weeks 3
Population: Data were not available for the calculations in the patients of 1 mg idursulfase-IT group at Week 3. Serum samples were not obtained from one patient in the 30mg Idursulfase-IT group at Week 3 after IV and IT administration.
Measure: Mean (Standard Deviation); unit: min*ng/mL
Groups:
- Idursulfase IT (1 mg): monthly using an intrathecal drug delivery device (IDDD.
Arm/Group | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 0 | 4 | 3
min*ng/mL |  | 140022 (45479) | 228840 (37909)

10. Secondary Outcome: Concentration of Idursulfase in Serum After Repeated Doses of Intrathecal Idursulfase-IT Given in Conjunction With Elaprase
Time Frame: Weeks 23
Population: Only 1 patient out of 4 in the 1mg dose yielded sufficient data to calculate AUC.
Measure: Mean (Standard Deviation); unit: min*ng/mL
Groups:
- Idursulfase IT (1 mg); Idursulfase IT (30 mg): monthly using an intrathecal drug delivery device (IDDD) Value represents concentration at 36 hours post drug administration.
- Idursulfase IT (10 mg): monthly using an intrathecal drug delivery device (IDDD) Value represents concentration at 24 hours post drug administration
Arm/Group | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 1 | 4 | 4
min*ng/mL | 31481 | 150544 (43871) | 174247 (49795)

11. Secondary Outcome: % Change From Baseline in Urinary GAG
Time Frame: Baseline to Week 27
Measure: Mean (Standard Error); unit: % Change
Groups:
- Control: Untreated Patients, Observed Value
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Number analyzed (Participants) | 4 | 4 | 4 | 4
% Change | -7.67 (20.820) | 37.83 (27.971) | -22.38 (4.840) | 29.70 (13.700)

ADVERSE EVENTS:
Time Frame: Time of informed consent until 30 days after the patients end of study visit.
Arm/Group | Control | Idursulfase IT (1 mg) | Idursulfase IT (10 mg) | Idursulfase IT (30 mg)
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/4 | 2/4 | 2/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=4) | Idursulfase IT (1 mg) (N=4) | Idursulfase IT (10 mg) (N=4) | Idursulfase IT (30 mg) (N=4)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) — Event considered possibly related to the device
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Event not related to investigational treatment or device
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Event not related to investigational treatment or device
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Complication of device insertion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Untreated control patients did not have IDDD implanted
Device breakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device connection issue (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=4) | Idursulfase IT (1 mg) (N=4) | Idursulfase IT (10 mg) (N=4) | Idursulfase IT (30 mg) (N=4)
Upper respiratory tract (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 4 (5)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anorectal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microcystosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pica (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal Behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Personality Change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staring (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (5)
Hyperreflexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pyramidal Tract Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory Integrative Dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle Ear Infusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motion Sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Atrial Hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left Ventricular Hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral Valve Prolapse (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Fluctuation (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (7) | 3 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (2) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toe Walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bicuspid Aortic Valve (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (3)
Catheter Related Complication (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Implant Site Swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Catheter Site Erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant Site Effusion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant Site Erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant Site Scar (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Odema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Diastolic Decreased (Investigations) | 0 (0) | 2 (6) | 3 (9) | 2 (10)
Blood Pressure Systolic Increased (Investigations) | 1 (1) | 2 (10) | 2 (5) | 2 (8)
Blood Pressure Systolic Decreased (Investigations) | 0 (0) | 1 (7) | 2 (3) | 2 (6)
Heart Rate Decreased (Investigations) | 1 (1) | 2 (8) | 1 (2) | 1 (1)
Blood Pressure Decreased (Investigations) | 0 (0) | 2 (4) | 2 (5) | 0 (0)
Blood Pressure Diastolic Increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 1 (5)
Protein Total Decreased (Investigations) | 0 (0) | 1 (1) | 2 (5) | 1 (1)
Body Temperature Decreased (Investigations) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
CSF Cell Count Increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (2)
CSF Protein Increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (2)
Cardiac Murmur (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Blood Chloride Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Body Temperature Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CSF Glucose Decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Red Blood Cells CSF Positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Calcium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Triglycerides Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CSF White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart Sounds Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mean cell volume abnormal (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PCO2 Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Rate Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Rate Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroxine Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 3 (3) | 4 (5) | 4 (7) | 2 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Agitation Post-Operative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns First Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication of Device Insertion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device Breakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device Connection Issue (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device Failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Drug Delivery System Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical Device Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suture Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic Lumbar Puncture (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Extractions (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Untreated control group were not implanted with IDDD. Concentration of idursulfase in all CSF samples post single dose of idursulfase-IT were below LLOQ(Lower limit of quantitation) of the bioanalytical method therefore no results are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information(excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.